CLINICAL TRIAL: NCT05143125
Title: Clinical Study of Decitabine Combined With NK Cell Infusion in the Treatment of Malignant Tumors
Brief Title: Treatment of Malignant Tumors With NK Cell
Acronym: NK cell
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HEM-ONCO-009
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-02

CONDITIONS: Malignancy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Decitabine combined with NK cell infusion as post-remission therapy
  Interventions: Biological: Decitabine combined with NK cell infusion

INTERVENTIONS:
Biological: Decitabine combined with NK cell infusion — Decitabine combined with NK cell infusion

SUMMARY:
Natural killer cells (NK cells) are derived from bone marrow lymphoid stem cells, which are a type of lymphocytes that can non-specifically kill tumor cells and virus-infected cells without pre-sensitization. NK cells can not only directly kill malignant diseased cells, but also participate in the regulation of immune cell response and play a role in a variety of tumor immunotherapy strategies. The 2-year survival rate of NK cells combined with stem cell therapy for patients with hematological malignancies reached 36%, which is significantly higher than the 2-year survival rate (about 15%) of stem cell therapy alone, which can extend the disease-free survival period of leukemia patients by an average of 1.5 years. Relapsed and refractory leukemia can achieve a complete remission rate of up to 40%.

DETAILED DESCRIPTION:
Natural killer cells (NK cells) are derived from bone marrow lymphoid stem cells, which are a type of lymphocytes that can non-specifically kill tumor cells and virus-infected cells without pre-sensitization. NK cells can not only directly kill malignant diseased cells, but also participate in the regulation of immune cell response and play a role in a variety of tumor immunotherapy strategies. The 2-year survival rate of NK cells combined with stem cell therapy for patients with hematological malignancies reached 36%, which is significantly higher than the 2-year survival rate (about 15%) of stem cell therapy alone, which can extend the disease-free survival period of leukemia patients by an average of 1.5 years. Relapsed and refractory leukemia can achieve a complete remission rate of up to 40%. However, NK cell therapy alone or the use of autologous NK cells to treat solid tumors is not effective. In clinical trials related to rectal cancer, esophageal cancer, kidney cancer, and gastric cancer, the clinical response of NK cell adoptive therapy is not good. A phase II clinical study found that the disease control rate of patients with ovarian cancer and breast cancer after radiotherapy and chemotherapy can reach about 60% by NK cell infusion. The main reason for the low treatment efficiency of solid tumors is related to the immunosuppressive effect of the tumor microenvironment. Combination therapy is a potential breakthrough. Researches targeting tumor immune microenvironment, targeting tumor cells and combined with NK cell therapy have shown tumor therapeutic potential. NK cells combined with IgG1 antibody treatment of gastric cancer and colon cancer in about 50% of patients with partial remission, and 17% of patients are in stable condition. In summary, the combined application of the demethylation drug DAC and NK cell infusion may be a new clinical strategy for the treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 (including 18 and 70 years old);
2. Those who have been diagnosed as malignant tumor by pathological and histological examination, have received anti-tumor treatment and are in remission;
3. The ECOG score of the patient is less than 2 points;
4. The patient did not receive any chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) and other anti-tumor treatments within 4 weeks before enrollment, and his previous treatment-related toxicity had returned to grade <1 (hair loss, peripheral nerves) at the time of enrollment Except for low-level toxicity such as inflammation);
5. The patient's intravenous access is unobstructed, which can meet the needs of intravenous drip;
6. The patient voluntarily participates and signs an informed consent form, and follows the research treatment plan and visit plan.

Exclusion Criteria:

1. The patients used high-dose hormones within 1 week before enrollment (except for patients using inhaled hormones);
2. People with severe autoimmune diseases, immunodeficiency diseases or severe allergies;
3. Patients who have been treated with other cellular immune products (DC, T, CTL, CAR-T, etc.);
4. The patient had an uncontrollable infection within 4 weeks before enrollment;
5. Active B HBV DNA>1000copy/mL/C virus hepatitis (anti-HCV positive, HCV RNA positive), HIV positive, syphilis positive;
6. The patient has participated in other clinical studies within 6 weeks before enrollment;
7. Patients suffering from mental illness;
8. The patient has drug abuse/addiction and medical, psychological or social conditions that may interfere with research or have an impact on the evaluation of research results;
9. The patient has alcohol dependence;
10. Women who are pregnant (positive urine/blood pregnancy studies) or breastfeeding; men or women who have a pregnancy plan within the past year; patients cannot be guaranteed to take effective contraceptive measures during the study period;
11. According to the judgment of the investigator, the patient has other conditions that are not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of initial treatment to the end of follow up, up to 2 years
  DFS

SECONDARY OUTCOMES:
Overall survival rate | From admission to the end of follow up, up to 2 years.
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No